CLINICAL TRIAL: NCT05976321
Title: An Open-Label, Phase 1 Study to Compare Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of TAK-279 in Subjects With or Without Hepatic Impairment
Brief Title: A Study of TAK-279 in Adults With or Without Liver Damage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-279-1004
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1, Moderate HI: TAK-279 50 mg (Experimental): Participants with moderate HI will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part A of the study.
  Interventions: Drug: TAK-279
- Cohort 2, Normal Hepatic Function: TAK-279 50 mg (Experimental): Participants with normal hepatic function will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part A of the study. Based on an evaluation of the results from Part A, additional participants with normal hepatic function may be enrolled in Part B of the study.
  Interventions: Drug: TAK-279
- Cohort 3, Mild/Severe HI: TAK-279 50 mg (Experimental): Participants with mild/severe HI will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part B of the study based on an evaluation of the results from Part A.
  Interventions: Drug: TAK-279

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsules.

SUMMARY:
The main aim of this study is to find out how the body processes 1 dose of TAK-279 (pharmacokinetics) in participants with liver problems compared to participants without liver problems. Other aims are to check for side effects from TAK-279 and to learn how well participants tolerate 1 dose of TAK-279.

The participants will need to stay at the clinic for 11 days.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. The study will assess the safety and tolerability of single oral dose of TAK-279 in participants with moderate (Part A) and mild or severe (Part B) hepatic impairment (HI) compared to healthy participants with normal hepatic function.

The study will enroll up to 32 participants. Participants will be assigned to following study arms:

* Cohort 1, Moderate HI: TAK-279 50 mg
* Cohort 2, Normal Hepatic Function: TAK-279 50 mg
* Cohort 3, Mild/Severe HI: TAK-279 50 mg

This multi-center trial will be conducted in the United States. The overall duration of the study is approximately 42 days. Participants will be followed up for 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

A. Participants with Hepatic Impairment:

The participants must fulfill the following inclusion criteria to be eligible for participation in the study (participants who do not qualify based on a reversible condition or mild intercurrent illness may be re-screened after the condition is resolved. Screening tests may be repeated if in the Investigator's opinion the test needs to be repeated):

1. Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.
2. Adult male or female participant aged ≥18 years, at screening.
3. Has a body weight greater than 50 kilograms (kg) and has a body mass index (BMI) ≥18.0 and ≤42.0 kilograms per meter square (kg/m^2), at screening.
4. Continuous non-smoker or moderate smoker (≤10 cigarettes/day or the equivalent [including electronic cigarettes]) before screening. Participant must agree to smoke no more than 5 cigarettes or equivalent/day (including electronic cigarettes) from the 7 days prior to TAK-279 dosing.
5. Aside from HI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, or screening clinical laboratory profiles, as deemed by the Investigator or designee, including:

   * Supine blood pressure (BP) is ≥90/40 millimeters of mercury (mmHg) and ≤150/95 mmHg, at screening.
   * Supine pulse rate (PR) is ≥40 beats per minute (bpm) and ≤99 bpm, at screening.
   * Estimated creatinine clearance (CrCl) ≥60 millilitres per minute (mL/min) (using Cockcroft-Gault formula) at screening. Both estimated CrCl and estimated glomerular filtration rate (eGFR) using modification of diet in renal disease (MDRD) formula will be reported.
6. Have had chronic HI for at least 3 months before screening, and the HI must be stable, i.e., no significant changes in hepatic function in the 30 days preceding screening (or since the last visit if within 3 months before screening).
7. Has a score on the Child-Pugh Class at screening as follows:

   * Severe HI cohort, Child-Pugh Class C: ≥10 and ≤15.
   * Moderate HI cohort, Child-Pugh Class B: ≥7 and ≤9.
   * Mild HI cohort, Child-Pugh Class A: ≥5 and ≤6.
8. Female participants of childbearing potential agree to comply with any acceptable contraceptive requirements of the protocol.

B. Healthy Participants:

1. Understands the study procedures in the ICF and be willing and able to comply with the protocol.
2. Adult male or female participant aged ≥18 years, at screening. Participant will be matched to a participant with HI by age (±10 years) and sex.
3. Has a body weight greater than 50 kg and has a BMI ≥18.0 and ≤42.0 kg/m^2, at screening. Participant will be matched a participant with HI by body weight (±15 kg).
4. Continuous non-smoker or moderate smoker (≤10 cigarettes/day or the equivalent [including electronic cigarettes]) before screening. Participant must agree to smoke no more than 5 cigarettes or equivalent/day (including electronic cigarettes) from the 7 days prior to TAK-279 dosing.
5. Medically healthy with no clinically significant medical history, physical examination, vital signs, or screening clinical laboratory profiles, as deemed by the Investigator or designee, including:

   * Supine BP is ≥90/40 mmHg and ≤150/95 mmHg, at screening.
   * Supine PR is ≥40 bpm and ≤99 bpm, at screening.
   * Liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and total bilirubin (TBILI) within the upper limit of normal (ULN) at screening and at check-in.
   * Estimated CrCl ≥60 mL/min (using Cockcroft-Gault formula) at screening. Both estimated CrCl and eGFR using MDRD formula will be reported.
6. Female participants of childbearing potential agree to comply with any acceptable contraceptive requirements of the protocol.

Exclusion Criteria:

A. Participants with Hepatic Impairment:

The participant must be excluded from participating in the study if the participant:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of screening or expected during the conduct of the study.
2. Has history or presence of clinically significant medical or psychiatric condition or disease (aside from HI) in the opinion of the Investigator or designee.
3. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to dosing, as assessed by the Investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to dosing.
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced within 60 days prior to dosing.
   * Opportunistic infections (e.g., Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   * Cancer or lymphoproliferative disease within 5 years prior to dosing, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix is not exclusionary.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
   * Liver or other solid organ transplant.
5. Has history or presence of alcoholism and/or drug abuse within the past 6 months prior to dosing, as determined by the Investigator or designee.
6. Has history or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
7. Female with a positive pregnancy test or who is lactating.
8. Has electrocardiogram (ECG) abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the study, in the opinion of the Investigator or designee.
9. Has positive results for the urine or saliva drug screen at screening or check-in, unless the positive drug screen is due to prescription drug use that is approved by the Investigator or designee and Sponsor.
10. Has positive results for urine or breath alcohol screen at screening or check-in.
11. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements).
12. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
13. Has made a donation of blood or had significant blood loss within 56 days prior to dosing.
14. Has made a plasma donation within 7 days prior to dosing.
15. Participated in another clinical study within 30 days prior to dosing. The 30-day window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
16. Herpes infections:

    * Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1.
    * Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes simplex virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
17. Positive results for non-herpetic viral diseases at screening:

    * Hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV Ribonucleic acid (RNA) (nucleic acid test or Polymerase chain reaction [PCR]).
    * Hepatitis B surface antigen (HBsAg)+, hepatitis B virus Deoxyribonucleic acid (DNA), or Hepatitis B core antibody (HBcAb)+ with positive hepatitis B virus DNA.
    * Human immunodeficiency virus (HIV).
18. Tuberculosis (TB):

    * Has history of active TB infection, regardless of treatment status.
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the Investigator or designee.
    * Has evidence of latent tuberculosis infection (LTBI) as evidenced by a positive QuantiFERON-TB Gold (QFT) result OR 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis. Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines).
    * Has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.
19. The participant has any of the following:

    * A history of esophageal or gastric variceal bleeding within the past 6 months and for which varices have not been adequately treated with medication and/or surgical procedure(s), or a history of bleeding due to gastric ulcers within the past 6 months, or presence of medium or large varices or varices with red wale signs based on a previous esophagogastroduodenoscopy (EGD) within 6 months before screening that have not been treated, if EGD performed within the past 6 months prior to screening is available.
    * The participant has grade >2 hepatic encephalopathy assessed using the West Haven criteria.
    * The participant has evidence of hepatopulmonary syndrome or portal-pulmonary hypertension.
    * The participant has portal vein thrombosis, transjugular intrahepatic portosystemic shunt, or surgical portosystemic shunt.
    * Severe ascites, except for participants in severe HI cohort, if the participant is medically stable, in the opinion of the Investigator or designee.
20. Participants with ALT or AST >5x ULN at screening, with a single repeat permitted to assess eligibility, if needed.

B. For Healthy Participants:

The participant must be excluded from participating in the study if the participant:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of screening or expected during the conduct of the study.
2. Has history or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to dosing, as assessed by the Investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to dosing.
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced within 60 days prior to dosing.
   * Opportunistic infections (e.g., Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   * Cancer or lymphoproliferative disease within 5 years prior to dosing, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix is not exclusionary.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
   * Liver or other solid organ transplant.
5. Has history or presence of alcoholism and/or drug abuse within the past 2 years prior to dosing, as determined by the Investigator or designee.
6. Has history or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
7. Female with a positive pregnancy test or who is lactating.
8. Has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the study, in the opinion of the Investigator or designee.
9. Has positive results for the urine or saliva drug screen at screening or check-in, unless the positive drug screen is due to prescription drug use that is approved by the Investigator or designee and Sponsor.
10. Has positive results for urine or breath alcohol screen at screening or check-in.
11. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements).
12. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
13. Has made a donation of blood or had significant blood loss within 56 days prior to dosing.
14. Has made a plasma donation within 7 days prior to dosing.
15. Participated in another clinical study within 30 days prior to dosing. The 30-day window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
16. Herpes infections:

    * Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1.
    * Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes simplex virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
17. Positive results for non-herpetic viral diseases at screening:

    * HCV antibody and a positive confirmatory test result for HCV RNA (nucleic acid test or PCR).
    * HBsAg+, hepatitis B virus DNA, or HBcAb+ with positive hepatitis B virus DNA.
    * HIV.
18. TB:

    * Has history of active TB infection, regardless of treatment status.
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the Investigator or designee.
    * Has evidence of LTBI as evidenced by a positive QFT result OR 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis. Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines).
    * Has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-279 | Predose and at multiple time points post dose from Days 1 to 10
AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-279 | Predose and at multiple time points post dose from Days 1 to 10
AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for TAK-279 | Predose and at multiple time points post dose from Days 1 to 10

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to 14 days
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Number of Participants With Adverse Events of Special Interest (AESIs) | Up to 14 days
Number of Participants With Clinically Significant Vital Signs | Up to 10 days
Number of Participants With Clinically Significant Electrocardiogram Findings | Up to 10 days
Number of Participants With Clinically Significant Laboratory Values | Up to 10 days
Number of Participants With Clinically Significant Physical Examination Findings | Up to 10 days
Cmax,u: Maximum Observed Unbound TAK-279 Plasma Concentration | Post dose at multiple timepoints from Day 1 to Day 2
AUClast,u: Area Under the Unbound Drug Concentration-time Curve, From Time 0 to the Last Quantifiable Concentration of TAK-279 | Post dose at multiple timepoints from Day 1 to Day 2
AUC∞,u: Area Under the Unbound Drug Concentration-time Curve, From Time 0 to Infinity of TAK-279 | Post dose at multiple timepoints from Day 1 to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/8db7580343404867?idFilter=%5B%22TAK-279-1004%22%5D